CLINICAL TRIAL: NCT00072137
Title: Phase I Study of Intravesical Recombinant Fowlpox - GM-CSF (rF-GM-CSF) and/or Recombinant Fowlpox-TRICOM (rF-TRICOM) in Patients With Bladder Carcinoma Scheduled for Cystectomy
Brief Title: Neoadjuvant Intravesical Vaccine Therapy in Treating Patients With Bladder Carcinoma Who Are Undergoing Cystectomy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00020; NCI-2009-00020 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000335473; 050301 (Other: Rutgers Cancer Institute of New Jersey); 5585 (Other: CTEP); U01CA132194 (NIH); P30CA072720 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Adenocarcinoma; Bladder Squamous Cell Carcinoma; Bladder Urothelial Carcinoma; Recurrent Bladder Carcinoma; Stage I Bladder Cancer; Stage II Bladder Cancer; Stage III Bladder Cancer; Stage IV Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

ARMS (3):
- Arm A (rf-GM-CSF, closed to accrual 10/2004) (Experimental): Patients receive recombinant fowlpox GM-CSF vaccine adjuvant intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.
  Interventions: Biological: Recombinant Fowlpox GM-CSF Vaccine Adjuvant; Procedure: Therapeutic Conventional Surgery; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis
- Arm B (rf-TRICOM, closed to accrual 10/2004) (Experimental): Patients receive recombinant fowlpox-TRICOM vaccine intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.
  Interventions: Biological: Recombinant Fowlpox-TRICOM Vaccine; Procedure: Therapeutic Conventional Surgery; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis
- Arm C (rfTRICOM and rf-GM-CSF) (Experimental): Patients receive recombinant fowlpox-TRICOM vaccine combined with recombinant fowlpox GM-CSF vaccine adjuvant intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.
  Interventions: Biological: Recombinant Fowlpox-TRICOM Vaccine; Biological: Recombinant Fowlpox GM-CSF Vaccine Adjuvant; Procedure: Therapeutic Conventional Surgery; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Recombinant Fowlpox-TRICOM Vaccine — Given intravesically
  Other Names: Recombinant Fowlpox-TRICOM; rF-TRICOM (B7.1.iCAM1-LFA3-Fowlpox)
  Arms: Arm B (rf-TRICOM, closed to accrual 10/2004); Arm C (rfTRICOM and rf-GM-CSF)
Biological: Recombinant Fowlpox GM-CSF Vaccine Adjuvant — Given intravesically
  Other Names: Fowlpox-Sargramostim; rF-GM-CSF; rF-Sargramostim
  Arms: Arm A (rf-GM-CSF, closed to accrual 10/2004); Arm C (rfTRICOM and rf-GM-CSF)
Procedure: Therapeutic Conventional Surgery — Undergo cystectomy
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of vaccine therapy given directly into the bladder in treating patients who are undergoing surgery to remove all or part of the bladder. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Giving a vaccine directly into the bladder before surgery may cause a stronger immune response and keep tumor cells from coming back after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of intravesical administration of recombinant fowlpox virus encoding three different costimulatory molecules (B7.1, ICAM-1,LFA-3) called TRICOM (-rF-TRICOM) (recombinant fowlpox-TRICOM vaccine) and/or recombinant fowlpox encoding sargramostim (GM-CSF) (rF-GM-CSF) (recombinant fowlpox GM-CSF vaccine adjuvant) in the treatment of patients with carcinoma of the bladder scheduled for cystectomy.

SECONDARY OBJECTIVES:

I. Determine the kinetics of viral infection and gene function as well as host response to intravesical recombinant fowlpox virus in the treatment of bladder cancer.

OUTLINE: This is a dose-escalation study. Patients are alternately assigned to Arms A and B. Once Arms A and B have finished accrual, patients are assigned to Arm C.

ARM A (closed to accrual 10/2004): Patients receive recombinant fowlpox GM-CSF vaccine adjuvant intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.

ARM B (closed to accrual 10/2004): Patients receive recombinant fowlpox-TRICOM vaccine intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.

ARM C: Patients receive recombinant fowlpox-TRICOM vaccine combined with recombinant fowlpox GM-CSF vaccine adjuvant intravesically over 2 hours for 4 weekly doses (on days 1, 8, 15, and 22) with the last dose given 4-6 days prior to cystectomy.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity. All patients undergo cystectomy 4-6 days following the last intravesical instillation.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically documented bladder cancer including: transitional cell carcinoma, adenocarcinoma, or squamous cell carcinoma including carcinoma in situ (CIS) requiring cystectomy as a standard therapy for his/her tumor stage and be scheduled for this surgical procedure; patients should not be candidates for neoadjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Estimated life expectancy 6 or more months
* Prior therapy with intravesical Bacille Calmette-Guerin (BCG) and/or chemotherapy is allowed; patient must be at least 2 months beyond the instillation of any prior intravesical agent; patients should not have received systemic chemotherapy, radiation therapy, immunotherapy or systemic doses of steroids for at least 4 weeks prior to starting vaccination and have recovered from all acute toxicities of previous treatment; patients who have received neoadjuvant chemotherapy or radiation therapy to the bladder will be ineligible for this study
* Serum creatinine < 1.5 mg/dl or a creatinine clearance > 60 ml/min
* Bilirubin < 2.0 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 x normal range
* Absolute neutrophil count (ANC) > 1500/mm^3
* Platelets > 75000/mm^3
* Patients must not have known immunodeficiency disorder (acquired immunodeficiency syndrome [AIDS], severe combined immunodeficiency [SCID], Wiskott-Aldrich syndrome, etc.); study candidates will not be specifically screened for these, unless clinically indicated; if indicated, the referring physician will do the evaluation
* No active/uncontrolled infections
* Pregnant women or nursing mothers are ineligible; women with reproductive potential must have negative pregnancy test and are prohibited from sexual intercourse during this study (while receiving vaccine and at least 1 month following last dose); sexual abstinence (as opposed to contraception only) is necessary; similarly, male patients also must avoid sex for the same period as above
* No uncontrolled psychiatric illness or medical illness that the principal investigator feels will compromise the patient's tolerance of the study treatment
* Patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines; patients who cannot provide informed consent will not be eligible for the study

Exclusion Criteria:

* Altered immune-competence:

  * Current or imminent steroid therapy or active antibiotic therapy (antibiotics given for prophylaxis are allowed)
  * Immune deficiency disease or immunosuppressive therapy in the patient
* Present or history of an autoimmune disease in the patient (e.g. autoimmune neutropenia, thrombocytopenia, or hemolytic anemia; systemic lupus erythematosus, Sjogren syndrome, or scleroderma; myasthenia gravis; Goodpasture syndrome; Addison's disease, Hashimoto's thyroiditis, active Graves' disease, or other diseases which qualify as autoimmune in origin)
* History of allergy to eggs as this vaccine is manufactured in chicken embryo cells
* Patients with any presence of liver function abnormalities, exposure to toxins, ongoing alcohol consumption, history of liver disease and/or history of hepatitis that may suggest persistent disease
* Any concurrent active second malignancy or any malignant tumor within the prior 5 years with the exception of a superficial squamous or basal cell skin carcinoma or in situ carcinoma of the cervix or prostate
* Pregnancy
* Patients with active ischemic heart disease (i.e. class III or IV cardiac disease-New York Heart Association), a recent history of myocardial infarction (within the last 6 months), history of congestive heart failure, ventricular arrhythmias or other arrhythmias requiring therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-10; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) assessed by Common Toxicity Criteria (CTC) | Up to 39 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weiss, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States